CLINICAL TRIAL: NCT05349058
Title: Assessment of Myocardial Injury in Patients Treated With Immune Checkpoint Inhibitors
Acronym: MIICI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Flinders University (Other)
Collaborators: Flinders Medical Centre (Other Government); Lyell McEwin Hospital (Other Government)
Responsible Party: Principal Investigator, Joseph Selvanayagam, Professor Joseph Selvanayagam, Flinders University
Other Study IDs: MIICI2022/1.3
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Myocarditis; Immune Checkpoint Inhibitors; Cardiotoxicity; Myocardial Injury
Keywords: Immune Checkpoint Inhibtors (ICI); Cardiotoxicity
MeSH Terms: conditions — Myocarditis; Cardiotoxicity | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICI patients: Patients receiving an Immune Checkpoint Inhibitor as treatment for their malignancy
  Interventions: Drug: Immune Checkpoint Inhibitors

INTERVENTIONS:
Drug: Immune Checkpoint Inhibitors — Patients receive Immune Checkpoint Inhibitor as per oncology protocol

SUMMARY:
ICI's have become the first-line treatment for patients with various malignancies. Although case studies represent fulminant myocarditis, there is uncertainty in prevalence of subclinical myocardial injury induced by ICI's.

In this prospective study, ICI treatment naïve patients with no significant prior cardiovascular history were enrolled. Primary outcome was the prevalence and severity of cardiac Troponin I (cTnI) at 6 weeks following ICI. Secondary outcomes were change in global longitudinal strain (GLS) and right ventricular free wall strain (RV FWS) measured by echocardiography, myocardial injury as assessed by cardiovascular magnetic resonance (CMR) and major adverse cardiac events (MACE). MACE defined as composite of cardiovascular mortality, heart failure, hemodynamically significant arrhythmias or heart block at 3 months.

DETAILED DESCRIPTION:
There has been an increasing recognition of the relationship between immune surveillance and tumour proliferation over the last four decades. One of the most important therapeutic advances as a result of this knowledge expansion has been the development of immunotherapies such as Immune Checkpoints Inhibitors (ICI) for the treatment of a variety of malignancies. ICI's stimulate an overproduction of cytotoxic T cells, which are capable of mounting an attack on cancerous cells. There are currently seven different ICI's approved by the US Food and Drug Administration (FDA) and used as commercially available therapeutics. With an increased usage of ICI's, there has been increased reports of Immune Related Adverse Effects (IRAE's) caused by autoreactive T cells, one of these being cardiac muscle inflammation, or myocarditis. Acute fulminant myocarditis can result in heart failure, cardiogenic shock and/or arrhythmias with a reported mortality rate of 25-56% within 3-10 years. Whilst ICI induced fulminant myocarditis is rare, little is known about the rates of subclinical myocardial injury and the cardiac functional and structural effects of ICI's over time.

Advanced cardiac imaging such as Cardiac Magnetic Resonance (CMR) and speckle tracking echocardiography (Echo) facilitate the early diagnosis of myocardial injury. CMR is non-invasive, free of ionizing radiation, highly sensitive and offers a variety of imaging parameters such as LGE, T1 mapping, T2 mapping to aid in myocardial tissue characterisation. Echo strain via speckle tracking echocardiography can depict early indications of cardiac dysfunction prior to the onset of functional changes, therefore abnormal strain measurements such as abnormal global longitudinal strain (GLS) and right ventricular free wall strain (RV FWS) occur prior to changes in left ventricular ejection fraction (LVEF). Cardiac biomarkers such as cardiac Troponin I (cTn I) and N-Terminal-Pro-hormone-B- type Natriuretic Peptide (NT-pro BNP) assess for myocardial injury and hemodynamic stress respectively within the myocardium. As the frequency of ICI's use increases as a cancer therapy, the concerns regarding cardiotoxicity are ever present and there is a lack of prospective data regarding this. The likelihood of pericardial and skeletal muscle inflammation resulting in cTn elevation has been raised as a distinct possibility. Hence, there is current clinical uncertainty in (a) the prevalence and severity of cTn elevation in the setting of ICI, (b) the functional and structural changes (if any) associated with the cTn elevation, and (c) the long-term cardiac clinical outcomes associated with the cTn elevation in patients receiving ICI therapy.

Hypotheses and Aims Our primary hypothesis was that patients receiving ICI therapy will demonstrate subclinical myocardial injury in the absence of cardiac symptoms as detected by elevations of cardiac troponin. Our secondary hypothesis was that patients demonstrating elevated CTnI would also demonstrate myocardial oedema and/or necrosis on CMR and impairments in Echo strain as detected by TTE. The primary outcome measure was the percentage of study patients who demonstrated cTnI above normal range at 6 weeks post treatment. Secondary outcome measures were to assess LV and RV global and regional dysfunction post ICI therapy via echocardiography, changes in NT-pro BNP, myocardial injury assessed by CMR 6 weeks post treatment and the MACE rate at 3 months. Patients were screened for participation in the study according to the inclusion/exclusion criteria.

Methodology Prior to treatment with ICI, patients have blood investigations and echocardiography at baseline. This was repeated at 6 weeks (+/- 1 week) with the inclusion of a possible CMR. Any cardiac event was noted within 3 months of treatment. A data record was stored and password protected. This information was shared with the attending oncologist and any adverse reaction/cardiac event was noted.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent will be obtained before any assessment is performed
* ≥ 18 years of age, male or female
* Patients planned for treatment with ICI (PD-1 and /or PD-L1) for malignancy
* Treatment naïve to ICI
* Asymptomatic cardiac status
* LVEF ≥55% by echocardiography during the screening period or within 6 months prior to study entry

Exclusion Criteria:

* Any prior echocardiographic measurement of LVEF <55%
* Prior diagnosis and treatment for cardiac disease (myocardial infarction or angina, cardiomyopathy / heart failure, valvular heart disease)
* Elevated NT-proBNP > 600 pg/ml (> 900 pg/ml in the presence of atrial fibrillation).
* Life expectancy of less than 6 months
* Severe respiratory diseases requiring long-term oxygen therapy
* Patients enrolled in another clinical trial
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a asymptomatic cardiac status planned for treatment with Immune Checkpoint Inhibitor (ICI) (PD-1 and /or PD-L1) as apart of their protocol for malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-01-17 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac Troponin I (cTn I) | 6 weeks
  Change in cTnI

SECONDARY OUTCOMES:
N-terminal prohormone brain natriuretic peptide (NT-ProBNP) | 6 weeks
  Change in NT-ProBNP
Global and regional left ventricular (LV) and right ventricular (RV) dysfunction | 6 weeks
  Changes in LV ejection fraction (LVEF), Global Longitudinal Strain (GLS), Right Ventricular Free Wall Strain (RV FWS)
Major Adverse Cardiac Event (MACE) | 3 months
  Any occurrence of MACE. Which can be defined as composite of cardiovascular mortality, heart failure, hemodynamically significant arrhythmias or heart block at 3 months
Myocardial injury (CMR) | 6 weeks
  Myocardial injury as assessed by cardiac MRI. The measurements of LGE, T1 and T2 mapping

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Selvanyagam, Md, PhD, Principal Investigator — Flinders Univeristy
Locations (1):
- Flinders Medical Centre, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
No data will be shared to others